CLINICAL TRIAL: NCT01062126
Title: Advanced Bradycardia Device Feature Utilization and Clinical Outcomes
Brief Title: BRADYCARE: Advanced Bradycardia Device Feature Utilization and Clinical Outcomes
Acronym: BRADYCARE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD525
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Pacemaker
Keywords: Pacemaker; Advanced Features; Clinical Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pacemaker technology is constantly evolving. In the past 10 years, numerous advancements have been made in pacemaker therapy, diagnostics and connectivity. These advancements include automated capture, automated sensing, patient alert functions, algorithms minimizing ventricular pacing, automatic mode switching in response to atrial tachyarrhythmia, rate responsive pacing, advanced diagnostic features, remote monitoring and radiofrequency (RF) technology. However, little information is available on how these new features are being utilized by physicians in the real world and how these features impact patient outcomes.

This observational study will gather data on the patients' presenting clinical status, indication for device implantation, utilization of advanced device features, device therapy choices, clinical management and outcomes in a general pacemaker population.

The primary aim of the study is to evaluate the usage of advanced features and diagnostics in patients with St. Jude Medical pacemakers. The secondary aim of the study is to learn more about the progressive clinical outcomes in the general pacemaker patient population. The tertiary aim of the study is to evaluate the correlation between the usage of advanced features in pacemaker patients and the patient's clinical outcomes.

DETAILED DESCRIPTION:
Evaluation of Device Features and Diagnostics

* Programmed parameters: Advanced pacemaker features (Autocapture, Auto sensitivity control (ASC), Ventricular Intrinsic Preference (VIP®), Patient Notifier, RF telemetry, and newer advanced features)
* Device and lead measurements
* Number of AT/AF, VT/VF, PMT and AMS episodes

Evaluation of Clinical Parameters

* Indication for device implantation
* Cardiac and arrhythmia history
* Cardiac drug utilization
* Cardiac events: incidence and onset of symptomatic atrial fibrillation (AF), onset of heart failure (HF), incidence and onset of angina, occurrence of myocardial infarction (MI), occurrence of transient ischemic attack (TIA)/ischemic stroke, and occurrence of hemorrhagic stroke
* Modified Specific Activity Scale (SAS)
* Intrinsic QRS duration
* Left ventricular ejection fraction (LVEF)
* Adverse events
* All-cause, cardiovascular and heart failure hospitalizations
* All-cause, cardiovascular and heart failure mortality

ELIGIBILITY:
Inclusion Criteria:

* Patient has a current indication for a single-chamber (SR) or dual-chamber (DR) pacemaker or CRT-P device.
* Patient is implanted with an SJM Accent™ SR/DR, Accent™ SR/DR RF, Anthem™ CRT-P, Anthem™ CRT-P RF, or newer SJM pacemaker device.
* Patient is geographically stable and willing to comply with the required follow-up schedule.
* Patient is not pregnant or planning to become pregnant.
* Patient is >18 years of age.

Exclusion Criteria:

* Patient's life expectancy is less than 12 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for standard Pacemaker indications
Sampling Method: Non-Probability Sample
Enrollment: 3389 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott (previously St. Jude Medical)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects Enrolled in the Study: Patients implanted with an SJM Accent SR/DR, Accent SR/DR RF, Anthem CRT-P, Anthem CRT-P RF, or newer SJM pacemaker device
Period: Overall Study
Arm/Group | All Subjects Enrolled in the Study
Started | 3389
Completed | 2856
Not Completed | 533
Not completed — Death | 209
Not completed — All Withdrawals | 324

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Enrolled in the Study: All subjects that were enrolled in the study.
Arm/Group | All Subjects Enrolled in the Study
Number analyzed (Participants) | 3389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 559
  >=65 years | 2830
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1546
  Male | 1843
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 185
  Not Hispanic or Latino | 3175
  Unknown or Not Reported | 29
Region of Enrollment [Number; unit: participants]
  United States | 3389
Primary Indication for Pacemaker Implant [Count of Participants; unit: Participants]
  Sinus Node Dysfunction | 2427
  AV Node Block | 754
  Syncope | 220
  Pacemaker Replacement | 329
  PAVE | 55
  Others | 20
Cardiovascular History [Count of Participants; unit: Participants]
  Coronary Artery Disease | 1361
  Angina | 156
  Myocardial Infarction | 204
  Heart Failure | 25
  Hypertension | 2668
Ejection Fraction [Mean (Standard Deviation); unit: % of blood leaving heart at contraction] | 56.8 (9.9)
Other Medical History [Count of Participants; unit: Participants]
  Pulmonary disease | 335
  Hepatic/Renal disease | 306
  Diabetes | 869
  Peripheral vascular disease | 240
Medications [Count of Participants; unit: Participants]
  ACE Inhibitors/ARBs | 1659
  Aldosterone inhibitors | 64
  Anti-coagulants | 1064
  Antiarrhythmics - Class I | 103
  Antiarrhythmics - Class III | 356
  Antiplatelet | 1833
  Beta Blockers | 1653
  Calcium channel blockers | 936
  Cardiac glycosides | 239
  Diuretics | 1172
  Nitrates | 360
  Other cardiac | 351
  Positive Ionotropics | 11
  Statins | 150
Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 130.1 (19.6)
Diastolic BP [Mean (Standard Deviation); unit: mm Hg] | 72.2 (11.3)
Heart Rate [Mean (Standard Deviation); unit: beats per min (bpm)] | 69.4 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate at 1-year Post-implant
Description: Complication rate and 95% confidence interval at 1-year post-implant
Time Frame: 12 months
Population: All subjects enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of enrolled subjects
Arm/Group | All Subjects Enrolled in the Study
Number analyzed (Participants) | 3389
percentage of enrolled subjects | 1.12 [0.8 to 1.5]

ADVERSE EVENTS:
Time Frame: Adverse events reported during the 1-year study.
Arm/Group | All Subjects Enrolled in the Study
All-Cause Mortality (participants affected / at risk) | 209/3389
Serious Adverse Events (participants affected / at risk) | 38/3389
Other Adverse Events (participants affected / at risk) | 17/3389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Enrolled in the Study (N=3389)
Lead dislodgement or migration (Product Issues) | 14 (15)
Infection (Infections and infestations) | 6 (6)
Elevated pacing thresholds (Product Issues) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bleeding/Hematoma (Gastrointestinal disorders) | 1 (1)
Diaphragmatic/Phrenic Nerve Stimulation (Product Issues) | 1 (1)
Dehisence (Injury, poisoning and procedural complications) | 1 (1)
Lead Malfunction (Product Issues) | 1 (1)
Lead fracture (Product Issues) | 4 (4)
Loss of capture (Product Issues) | 1 (1)
Mid-sternal pain at the location of RA and RV leads (Injury, poisoning and procedural complications) | 2 (2)
Open wound at PG incision site (Injury, poisoning and procedural complications) | 1 (1)
Oversensing (Product Issues) | 1 (1)
Pericardial effusion (Injury, poisoning and procedural complications) | 2 (2)
Pericardial tamponade (Injury, poisoning and procedural complications) | 1 (1)
Pocket Revision- not Healing (Injury, poisoning and procedural complications) | 1 (1)
Set Screw not secured at Implant (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Enrolled in the Study (N=3389)
Elevated pacing thresholds (Product Issues) | 6 (6)
Oversensing (Product Issues) | 3 (3)
Atrial Arrhythmia (Cardiac disorders) | 2 (2)
Inappropriate device interaction (Product Issues) | 2 (2)
Loss of capture (Product Issues) | 2 (2)
Syncope (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days